CLINICAL TRIAL: NCT01217255
Title: Comparing the Burden of Illness of Hemophilia in the Developing and the Developed World: The Sao Paulo - Toronto Hemophilia Study
Brief Title: Comparing the Burden of Illness of Hemophilia in the Developing and the Developed World
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Brian Feldman, Division Head, Rheumatology, The Hospital for Sick Children
Other Study IDs: 1000020214
Record Dates: First submitted 2010-10-06; First posted 2010-10-08 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Hemophilia A; Hemophilia B
Keywords: Hemophilia; Burden of Illness; Pediatric; Quality of Life; Disability; Participation
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Brazilian Subject's: Subject's will be recruited from the Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paolo (HCFMUSP); Universidade Estadual de Campinas (UNICAMP); Universidade Federal de São Paulo (UNIFESP)
- Canadian Subject's: Recruited from The Hospital for Sick Children

SUMMARY:
Because of high cost, persons with hemophilia in many developing countries cannot afford adequate treatment. For example, many persons with hemophilia in India and China are only rarely treated with factor replacement in response to bleeds, and as a result many have developed significant arthropathy and disability. A pilot study in China estimated the mean Hemophilia Joint Health Score (HJHS) at 13.1 (SD 9.03) suggesting that these children had highly prevalent, severe joint disease. The lack of relationship between the HJHS and treatment history suggests overall inadequate therapy.

The proposed study will quantify the burden of arthropathy, physical disability, and quality of life (QoL) in boys with hemophilia in Brazil - where comprehensive treatment is just beginning to be widely available. This study will also provide an opportunity to compare these outcomes to those observed in Canada, where the dominant therapy has become life-long prophylaxis.

DETAILED DESCRIPTION:
In order to quantify the burden of illness in hemophilia, and to study the response to different treatments, it is necessary to have quantitative outcome measures of high validity and reliability. The International Prophylaxis Study Group (IPSG - chair Dr. Victor Blanchette) was established in 2001 with the stated purpose of developing and testing outcome tools for this purpose. The group has developed a magnetic resonance imaging (MRI) score for quantifying arthropathy (representing the domain of structure and function domain in the ICF framework), a quantitative physical examination score, and the Hemophilia Joint Health Score or HJHS, to replace the older and less sensitive World Federation of Hemophilia (WFH) score (representing the domain of structure and function in the ICF). In addition Canadian investigators have also developed a quality of life measure for boys with hemophilia, the Canadian Hemophilia Outcomes Kids' Life Assessment Tool or CHO-KLAT (representing the domain of participation in the ICF).

We will use these tools, and other validated measures, to begin to determine the burden of hemophilia in Brazil and compare it to the burden of disease in Canada. Additionally, we will use this study to demonstrate the validity of these tools in the Brazilian population.

ELIGIBILITY:
Inclusion criteria

* Hemophilia A or B moderate or severe as determined by serum factor activity ≤ 5%
* Age 7 - 18 yrs. inclusive
* At least one parent or guardian fluent in written Portuguese or English and able to complete the study outcome questionnaires.

Exclusion criteria

* None (Children with inhibitors will be allowed into the study for 2 reasons: i) our study aims to document the health of persons with hemophilia in a generalizable way, ii) not all children will have had inhibitor testing done.)

Ages: 7 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants will be a representative (random) sample of individuals from the comprehensive hemophilia treatment centres at HCFMUSP and SickKids. Boys between the ages of 7 and 18 years (inclusive) will be identified from the clinic ledgers at each of the centres. Using a computer generated random number list, proportionately stratified for Hemophilia A and B, and for moderate and severe disease (based on the baseline clinic proportions)
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2010-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Burden of Illness | 3 years
  Burden of disability for Brazilian and Canadian children will be be determined by analysis of the following domains:
  Structure and Function Domain (HJHS score, Biometrics,Radiographs) Activity Domain (ASK and FISH scales) Participation Domain (CHO-KLAT and PedsQL Quality of Life Questionnaire) Health Condition Domain (bleeding frequency) Personal Factors Domain (Ethnicity, level of education of parent/guardian, habitual exercise) Environmental Domain (Household income of parent/guardian)

SECONDARY OUTCOMES:
The Activity Scale for Kids (ASK) | Day 1
  Children's self-reported activities will be measured with the Activity Scales for Kids (ASK) as part of the Activity Domain
Functional Independence Scale for Hemophilia (FISH) | Day 1
  Observed activity limitations will be measured with the FISH as part of the Activity Domain.
  The FISH has been validated for use in developing countries. It consists of observed activities of daily living that are scored for quality.
Hemophilia Joint Health Score (HJHS) | Day 1
  The HJHS is a valid and reliable scored measure of joint structural limitations as applied to the index joints.
  This score will be a measure of the Structure and function domain.
Radiographs | Day 1
  Radiographs will be taken of all 6 index joints. This will be done as part of the structure and function domain.
Canadian Haemophilia Outcomes - Kids Life Assessment Tool (CHO-KLAT) | Day 1
  After the completion of the pre-study cultural validation of the Brazilian translation of the CHO-KLAT scale, we will use it as a Quality of Life tool to measure the Participation domain
Bleeding Frequency | Day 1
  Families will be interviewed to determine bleeding frequency in the last 6 months. This factor will be incorporated into the Health condition domain.
Biometrics | Days 1
  The height and weight will be compared to national nomograms.
Personal Factors | Day 1
  Ethnicity, level of education of the parent-guardian will be self-reported.
Environmental domain | Day 1
  Whether a subject lives in a rural or urban area and household income will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Brain M. Feldman, MD,MSc,FRCPC, Principal Investigator — The Hospital for Sick Children
Locations (4):
- Brazil (3):
  - Universidade Estadual de Campinas, UNICAMP, Campinas, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo, São Paulo
  - Universidade Federal de São Paulo (UNIFESP), São Paulo
- The Hospital for Sick Children, Toronto, Ontario, Canada